CLINICAL TRIAL: NCT06475950
Title: Impact of the "Kid'EM App" Digital Guidance Tool for Setting Rehabilitation Goals by the Rehabilitation Professional for Children with Chronic Conditions Impacting Physical Health (READ'APP'T)
Acronym: READ'APP'T
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 29BRC22.0257
Record Dates: First submitted 2023-07-28; First posted 2024-06-26 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-02

CONDITIONS: Children with Chronic Illnesses Affecting Physical Health
Keywords: Chronic disease; Children
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: "Kid'EM app" experimental group
  Rehabilitation professionals have access to the Kid'EM app tool, which guides them in setting goals.
  The app offers functionalities, including the selection of avatars by children, the identification of children's tastes and needs, the definition of SMART objectives, and the setting up of exchange spaces with parents and other professionals.
  The application enables the identification of environmental elements that may impact on the child's progress, and provides a note-taking space for the professional.
  Kidem app control group
  Rehabilitation professionals have access to a control application which has the same design, but does not offer guidance or a space for exchange with parents.
  The functionalities of the control application include the creation of the professional's account, selecting the child's pathology, identifying the child's tastes, and entering objectives without guidance.
  Professionals use their usual strategy to set goals."
Masking Description: The process of setting rehabilitation goals with "Kid'EM app" requires collaboration between the professional, the child and the family, preventing rehabilitation professionals and children and their families from being blindsided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kid'EM app" experimental group (Active Comparator): This group uses the Kid'EM app, which guides rehabilitation professionals in setting goals for each child. The app offers a variety of features, including the creation of patient accounts and records, identification of the child's likes and needs, definition of SMART goals, and spaces for exchanges with parents and other professionals. Parents also have access to the application.
  Interventions: Other: Kid'EM app" experimental group
- Kidem app control group (Sham Comparator): This group uses a control app that offers no guidance or space for exchange with parents. Professionals use their usual strategy to set goals. The functionalities of the control app are more limited, focusing on creating the professional's account, filling in the first letter of the child's first and last name, selecting the child's pathology, identifying the child's tastes, and filling in the objectives without guidance.
  Interventions: Other: Kid'EM app control group

INTERVENTIONS:
Other: Kid'EM app" experimental group — In the "Kid'EM app" experimental group arm, only the application used differs. Visits are organized in the same way as in the controle app arm.
  Visit 0 (Inclusion) + Visit 1 (V1) : Physical visit
  Children are included in the study by the investigator, formalized by signing a consent form.
  Parents fill in questionnaires
  Visit 2 (when 1st objective is set):
  Telephone interview to assess performance and satisfaction levels after the first goal has been set.
  Visit 3 (when setting the 2nd goal):
  Telephone interview to assess performance and satisfaction levels after the second goal has been set.
  Visit 4 (week 14 - end of study): Physical visit
  The questionnaires are again completed by the parents, either directly on a tablet or on paper for later input.
  Visit 4 bis:
  Telephone interview to assess performance and satisfaction levels after the work on the first two objectives.
  Visit 5 (focus group, optional post-study visit)
  Arms: Kid'EM app" experimental group
Other: Kid'EM app control group — Use of control application without guidance for goal setting
  Visit 0 (Inclusion) + Visit 1 (V1) : Physical visit
  Children are included in the study by the investigator, formalized by signing a consent form.
  Parents fill in questionnaires
  Visit 2 (when 1st objective is set):
  Telephone interview to assess performance and satisfaction levels after the first goal has been set.
  Visit 3 (when setting the 2nd goal):
  Telephone interview to assess performance and satisfaction levels after the second goal has been set.
  Visit 4 (week 14 - end of study): Physical visit
  The questionnaires are again completed by the parents, either directly on a tablet or on paper for later input.
  Visit 4 bis:
  Telephone interview to assess performance and satisfaction levels after the work on the first two objectives.
  Visit 5 (focus group, optional post-study visit)
  Arms: Kidem app control group

SUMMARY:
On an individual level, the first expected benefit for the child using the "Kid'EM app" would be an improvement in the quality of his or her rehabilitation goals, which would be more Specific, Measurable, Activity-related, Realistic and Time-defined (SMART). A second expected benefit for the child, thanks to the work carried out in rehabilitation sessions on objectives adapted to his or her needs and day-to-day life, encouraging commitment and motivation, would be to improve the effectiveness of the care offered to him or her, thereby enhancing autonomy and physical health. For parents, taking part in goal-setting, by contributing their knowledge of their child and his or her daily life, would increase their involvement in their child's care and improve their satisfaction with the care offered. By setting SMART functional goals and facilitating communication between therapist, child and family, we expect to see a more child- and family-centred approach to care.

On a collective level, the "Kid'EM app" proposal would, as recommended by the WHO, improve professional rehabilitation practices and facilitate convergence towards good clinical practices for professionals (physiotherapists, occupational therapists, PRMs, etc.), thereby increasing the efficiency of the child rehabilitation care system.

If its value is demonstrated, the Kid'EM app could be adapted for children with other chronic illnesses requiring non-motor rehabilitation follow-up. The digitization of this goal-setting tool means that this low-cost practice could be widely disseminated.

ELIGIBILITY:
Inclusion Criteria:

* Children with chronic illnesses affecting their physical health (e.g. Cerebral Palsy, Neuromuscular Disease, Brachial Plexus Paralysis, etc.).
* Children receiving rehabilitation care to promote autonomy and physical health.
* Child with at least one rehabilitation session/week with the same professional for a period of 3 months
* Children aged 5 to 17 wishing to participate in the study
* Parental consent for study participation and signature of consent form

Exclusion Criteria:

* Children without chronic illnesses that do not affect their physical health
* Children unable to express their views and priorities
* Children unable to collaborate with the rehabilitation professional when using the Kid'EM app
* Children already familiar with the "Kid'EM app" product
* Children whose parents are minors or unable to give informed consent

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Quality of the first two objectives set for each child during the 12-week 'Kid'EM app' or 'app control' period | Up to 3 weeks
  Quality, adequate or not (binary criterion, measured with the SMART goal evaluation method: SMART GEM), of the first two goals set for each child during the 12-week period of use of the "Kid'EM app" or "control app".
Quality of the first two objectives set for each child during the 12-week 'Kid'EM app' or 'app control' period | From week 14 to week 16
  Quality, adequate or not (binary criterion, measured with the SMART goal evaluation method: SMART GEM), of the first two goals set for each child during the 12-week period of use of the "Kid'EM app" or "control app".

SECONDARY OUTCOMES:
Evaluate the evolution of the child's satisfaction with rehabilitation care | Baseline
  - Evaluation of changes in satisfaction with the care offered to the child using an EVA scale completed by the children at V1.
Evaluate the evolution of the child's satisfaction with rehabilitation care | Week 14
  - Evaluation of changes in satisfaction with the care offered to the child using an EVA scale completed by the children at V4
Evaluation of the improvement in the child's family's satisfaction with rehabilitation care | Baseline
  Assessment of changes in satisfaction with the care offered to the child and his/her family using the CSQ8 scale completed by parents at V1.
Evaluation of the improvement in the child's family's satisfaction with rehabilitation care | Week 14
  Assessment of changes in satisfaction with the care offered to the child and his/her family using the CSQ8 scale completed by parents at V1.
Evaluation of the improvement in the effectiveness of care offered to children with chronic illnesses impacting physical health | Baseline
  - Evaluation of the evolution of the PEDI-CAT scale
Evaluation of the improvement in the effectiveness of care offered to children with chronic illnesses impacting physical health | Week 14
  - Evaluation of the evolution of the PEDI-CAT scale
Evaluation of the improvement in the effectiveness of care offered to children with chronic illnesses impacting physical health | Baseline
  - Evaluation of Disability Inventory-Computer Adaptative Test) completed by parents at V1.
Evaluation of the improvement in the effectiveness of care offered to children with chronic illnesses impacting physical health | Week 14
  - Evaluation of Disability Inventory-Computer Adaptative Test) completed by parents at V1.
Evaluation of the improvement in the effectiveness of care offered to children with chronic illnesses impacting physical health | Up to 3 weeks
  - Evaluation of the evolution of performance and satisfaction levels in achieving the first two rehabilitation goals determined by the rehabilitation professional, by parents at V2 (1st goal), using the CORM (Canadian Measure of Occupational Performance) evaluation methodology.
Evaluation of the improvement in the effectiveness of care offered to children with chronic illnesses impacting physical health | Up to 3 weeks
  - Evaluation of the evolution of performance and satisfaction levels in achieving the first two rehabilitation goals determined by the rehabilitation professional, by parents at V3 (2d goal), using the CORM (Canadian Measure of Occupational Performance) evaluation methodology.
Evaluation of the improvement in the effectiveness of care offered to children with chronic illnesses impacting physical health | Week 14
  - Evaluation of the evolution of performance and satisfaction levels in achieving the first two rehabilitation goals determined by the rehabilitation professional, by parents at V4 (both 1st goals), using the CORM (Canadian Measure of Occupational Performance) evaluation methodology.
Assessing how to improve the quality of care by promoting child- and family-centered care; | Baseline
  - Evaluation of the evolution of the MPOC (Measure of Processes Of Care) questionnaire completed by parents at V1.
Assessing how to improve the quality of care by promoting child- and family-centered care; | Baseline
  - Evaluation of the evolution of the MPOC (Measure of Processes Of Care) questionnaire completed by parents at V4.
Assessing how to improve the quality of care by promoting child- and family-centered care; | Baseline
  - Evaluation of the evolution of the MPOC SP (Measure of Processes Of Care Service Providers) questionnaire completed by rehabilitation professionals at V1
Assessing how to improve the quality of care by promoting child- and family-centered care; | Week 14
  - Evaluation of the evolution of the MPOC SP (Measure of Processes Of Care Service Providers) questionnaire completed by rehabilitation professionals at V4
Evaluation of parents' empowerment during child rehabilitation follow-up | Baseline
  - Assessment of changes in the Psychological Empowerment Scale (PES) completed by parents at V1
Evaluation of parents' empowerment during child rehabilitation follow-up | Week 14
  - Assessment of changes in the Psychological Empowerment Scale (PES) completed by parents at V4
Evaluation of the acceptability, usability and quality of the "Kid'EM app" | Week 14
  - Usability of the "Kid'EM app" application with the System Usability Scale (SUS) questionnaire by parents at V4 in the "Kid'EM app" group.
Evaluation of the acceptability, usability and quality of the "Kid'EM app" | Week 14
  - Quality of the "Kid'EM app" with the Mobile Application Rating Scale (MARS) by parents at V4 in the "Kid'EM app" group.
Evaluation of quality improvement in goal setting | From week 14 to week 16
  - Evaluation of the average SMART GEM score for the first two objectives established for each child during the 12-week period of use of the "Kid'EM app" or "control app".

CONTACTS AND LOCATIONS:
Locations (36):
- France (36):
  - Ildys Ty Yann, Angers
  - Les Capucins Angers, Angers
  - IEM Galaxie, Argeles
  - SESSAD 93 - Aulnay, Aulnay-sous-Bois
  - SESSAD APF Basse Goulaine, Basse-Goulaine
  - SMR Concarneau, Concarneau
  - Dispositif sensoriel et moteur Clos Chauveau - DIJON, Dijon
  - Sessad APF France Handicap du Finistère, Gouesnou
  - CAMSP APF Grenoble, Grenoble
  - Cabinet de Kinésithérapie - Elodie CREACH, Landerneau
  - SESSAD 93-Raincy, Le Raincy
  - Cabinet d'Ergothérapie - Maison des Korrigans, Lesneven
  - SESSAD A Denn Askell - KERPAPE, Lorient
  - CAMSP Nelson Mandela, Lyon
  - CAPEDIA, Lyon
  - CMCR Les Massues, Lyon
  - CMRP Romans Ferrari - Service Brulologie, Miribel
  - CMRP Romans Ferrari - Service Neurologie, Miribel
  - IEM La Marrière, Nantes
  - CHU Carémeau, Nîmes
  - Cabinet Jaures Kiné, Nîmes
  - Cabinet Sophie CHAPELLIER, Nîmes
  - IEM La Cigale, Nîmes
  - SESSAD La Cigale, Nîmes
  - IEM Ar Menn, Ploemeur
  - Centre Paul DOTTIN, Ramonville-Saint-Agne
  - SESSAD Henri Matisse, Rennes
  - SESSAD Romans, Romans-sur-Isère
  - SMR pédiatrique ILDYS, Roscoff
  - SESSAD Saint Etienne, Saint-Etienne
  - CHU Saint Etienne - MPR Pédiatrique, Saint-Etienne
  - CMPR Côte d'Amour, Saint-Nazaire
  - Centre de l'Arche, Saint-Saturnin
  - UGECAM Strasbourg, Strasbourg
  - SMR Vannes - Centre hospitalier bretagne atlantique, Vannes
  - Sessad Apf Voiron, Voiron

IPD SHARING:
Plan to Share IPD: Undecided